CLINICAL TRIAL: NCT05445830
Title: Physiological Characterization of Functional Limitations and Exercise Intolerance in Post-COVID Patients
Brief Title: Exercise Intolerance in Post-COVID Patients
Acronym: EXILE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Tommy Lundberg, Lecturer, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2021-05758-01
Record Dates: First submitted 2022-07-02; First posted 2022-07-06 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Post-COVID Syndrome
Keywords: Exercise intolerance; Acute exercise; Skeletal muscle; Cardiorespiratory fitness; Post-COVID syndrome
MeSH Terms: interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Upon collection, data will be pseudonymized (both group and intervention) to facilitate unbiased analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-covid patients (Experimental)
  Interventions: Procedure: High-Intensity-Interval-Exercise; Procedure: Moderate-Intensity-Continuous-Exercise; Procedure: Strength training; Procedure: Baseline assessment; Procedure: 1 year follow-up
- Control (Experimental)
  Interventions: Procedure: High-Intensity-Interval-Exercise; Procedure: Moderate-Intensity-Continuous-Exercise; Procedure: Strength training; Procedure: Baseline assessment; Procedure: 1 year follow-up

INTERVENTIONS:
Procedure: High-Intensity-Interval-Exercise — Subjects will perform high-intensity-interval exercise, where the acute exercise responses will be closely monitored, including measurements of O2 saturation, heart rate, blood pressure, borg scale and blood lactate. In addition, symptoms via multiple validated questionnaries and blood samples will be collected before, immediately after each exercise session to describe leukocyte and cytokine release as well as systemic metabolism. After a 48-hour rest period subjects will return to the laboratory for symptom assessment, submaximal exercise response (CPET), and blood sampling.
  Other Names: HIIE
Procedure: Moderate-Intensity-Continuous-Exercise — Subjects will perform moderate intensity continuous exercise, where the acute exercise responses will be closely monitored, including measurements of O2 saturation, heart rate, blood pressure, borg scale and blood lactate. In addition, symptoms via multiple validated questionnaries and blood samples will be collected before, immediately after each exercise session to describe leukocyte and cytokine release as well as systemic metabolism. After a 48-hour rest period subjects will return to the laboratory for symptom assessment, submaximal exercise response (CPET), and blood sampling.
  Other Names: MICE
Procedure: Strength training — Subjects will perform a series of a whole-body resistance exercises, where the acute exercise responses will be closely monitored, including measurements of O2 saturation, heart rate, blood pressure, borg scale and blood lactate. In addition, symptoms via multiple validated questionnaries and blood samples will be collected before, immediately after each exercise session to describe leukocyte and cytokine release as well as systemic metabolism. After a 48-hour rest period subjects will return to the laboratory for symptom assessment, submaximal exercise response (CPET), and blood sampling.
  Other Names: Resistance training
Procedure: Baseline assessment — Subjects will perform a series of baseline assessment including neurophysiological function, circulatory and vascular function, blood volume assessment, respiratory/ventilatory function, maximal oxygen uptake, strength, physical function and fitness, blood status and muscle biopsy.
Procedure: 1 year follow-up — Subjects will perform the same series of baseline assessment in 1-year time, including neurophysiological function, circulatory and vascular function, blood volume assessment, respiratory/ventilatory function, maximal oxygen uptake, strength, physical function and fitness, blood status and muscle biopsy.

SUMMARY:
The post-COVID syndrome poses an unprecedented challenge to modern society, affecting millions of people worldwide. Persistent fatigue and exercise intolerance are among the most common complaints of these subjects. The mechanisms of exercise intolerance in post-COVID subjects are remained yet unknown, which make the rehabilitation efforts complex and challenging. The overall goals of this project are to: 1) improve physiological understanding of symptoms in this clinical condition, 2) elucidate plausible mechanisms to explain exercise intolerance/symptom exacerbation, and finally 3) provide knowledge that can be directly applied in the clinical setting to improve diagnosis, care, and individualized rehabilitation of subjects with post-COVID syndrome. Post-COVID subjects and age/sex matched healthy controls will undertake a comprehensive set of physiological and functional assessments, followed by 3 experimental visits (in a randomized order), where acute exercise responses will be assessed in either continuous moderate intensity aerobic exercise, high intensity interval exercise, or strength training. The same set of physiological assessments will also be performed after 1 year in both post-COVID subjects and healthy-matched controls to better understand the time course of the syndrome. It is hypothesized that the mechanism responsible for exercise intolerance is linked to specific symptoms and will vary across subjects. However, it is expected that most post-COVID subjects will respond well to at least one type of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Verified test of covid-19 infection (PCR, or antigen or antibody before vaccination) (mandatory only for post-COVID group)
* Symptoms persisting for at least 3 months (validaded with DSQ-PEM questionnarie) (only for post-COVID group)

Exclusion Criteria:

* Subject's complaints may have been present before March 2020
* Previous history cardiovascular, respiratory disease or other autoimmune disease
* History of general anxiety syndrome or somatic symptom disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-exertional malaise (PEM) symptoms of post-COVID subjects and age/sex matched controls in response to different exercise trials. | Three exercises trials & 48 hours follow-ups of each trial
  Visual analog scale (VAS) 0-10 for 10 symptoms (fatigue, muscle pain, joint pain, memory, concentration, fever, sore throat, lymph nodes, headache, chills) will be used to assess symptoms exaggeration in response to 3 different exercise trials (high intensity interval training, moderate intensity continuous exercise and strength exercise) between the post-COVID subjects and age/sex matched controls.
  0=no pain/symptom to 10=maximal pain/symptom
  2 groups x 3 exercise sessions x 3 timepoints per exercise (pre, post and 48h post)

SECONDARY OUTCOMES:
Absolute immune cell count in blood samples of post-COVID subjects and age/sex matched controls in response to different exercise trials. | Three exercises trials & 48 hours follow-ups of each exercise trial
  Absolute immune count will be assessed via BD TruCount in collected blood samples (before, immediately-, and 48h-post) in response to different exercise trials (high intensity interval training, moderate intensity continuous exercise and strength exercise) across the post-COVID subjects and age/sex matched controls. PBMCs will be analysed for distribution of B cells, NK cells, monocytes, CD4+ T cells, CD8+ T cells, with additional panels to capture plasma, effector and memory cells.
Exploratory metabolomic and cytokine profiling using blood samples of post-COVID subjects and age/sex matched controls in response to different exercise trials. | Three exercises trials & 48 hours follow-ups of each exercise trial
  Metabolomic and cytokine profiling will be explored in collected blood samples (before, immediately-, and 48h-post) in response to different exercise trials (high intensity interval training, moderate intensity continuous exercise and strength exercise) across the post-COVID subjects and age/sex matched controls. Olink PEA platform and GC-MS at the Swedish Metabolomics Centre in Umea will be used and targeted analysis will include IL-6, TNF-a and IFN-g profiling.
Cardiac function in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Routine echocardiography wiil be performed to assess normal/abnormal heart structure and function in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up. A blinded observer will then quantify cardiac chamber dimensions and volumes, as well as the assessment of left ventricular systolic and diastolic function.
Respiratory function in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Routine spirometry wiil be performed to assess normal/abnormal lung structure and function in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up. The spirometry variables will be the forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), FEV% (FEV1/ VC MAX), maximum vital capacity (VC MAX), total lung capacity (TLC), and diffusing capacity of the lungs for carbon monoxide single breath corrected for Hb (DLCOc SB).
Arterial stiffness in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Non-invasive measurement of arterial stiffness via arteriography (Tensiomed) will be performed in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up. Higher pulse wave velocity (PWV) reflects higher degree of arterial stifness.
Dysautonomia in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Head-up TILT test (HUTT) will be performed according to clinical guidelines to assess normal or abnormal autonomic nervous system regulation in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up. Specifically, hemodynamic measurements (systolic blood pressure, diastolic blood pressure and heart rate) will be measured non-invasively using NOVA software at supine position and at standing. Medical doctor will then classify the patients as follows:
  1. Normal orthostatic reaction
  2. Post-orthostatic tachycardia syndrome (POTS): development of symptoms with a sustained heart rate increase of ≥ 30 bpm or ≥ 120 bpm within 10 minutes of standing, with no significant blood pressure difference, i.e., SBP decreased by ≥ 20mmHg and DBP ≥ 10mmHg
  3. Syncope: significant fall of HR or BP with loss of consciousness or inability to maintain posture
  4. Orthostatic hypotension: any HR increase with SBP decrease of ≥ 20mmHG or DBP decrease of ≥ 10mmHG
6-min walk test the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  The standard 6-min walk test will be performed to assess the physical function, including aerobic capacity in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up. Higher distance (in meters) covered by the participants reflects better physical function and aerobic capacity.
Handgrip strength the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  The gold standard Jama hydraulic hand dynamometer will be used to measure handgrip strength of the domiant hand to assess upper body muscular strength in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up.
Blood volume in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  The optimized carbon monoxide rebreathing method will be used to determine total hemoglobin, from which blood volume and plasma volume will later calculate using hemoglobin concentration [Hb] and hematocrit (Hct). This method will be conducted in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up.
Lower body muscle strength the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Maximal isometric (120°/s) and isokinetic strength (60°/s and 210°/s) will be measured using Biodex isokinetic dynamometer to assess lower body muscular strength in the post-COVID subjects and age/sex matched controls at baseline and 1y follow-up.
Nerve conduction studies the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Nerve conductions studies (NCS) will be conducted in the dominant lower and upper limb using the Cadwell Sierra Summit EMG system (Cadwell Industries, Inc., Kennewick, WA). Motor studies included the median, ulnar, fibular, and tibial nerves, and the compound muscle action potential (CMAP), distal latency (DL), conduction velocity (CV), and minimum F-wave latency will be recorded for all nerves. Sensory studies will include median, ulnar, radial, sural, and fibular nerves, and the sensory nerve action potential (SNAP) and CV will be recorded for all nerves. NCS will be performed in the post-COVID patients and age/sex matched controls at baseline and 1y follow-up
Needle Electromyography in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Needle electromyography (EMG) of 6 muscles (deltoid, biceps brachii, trapezius, anterior tibial, vastus medialis, and adductor magnus) will be performed using Sierra Summit EMG system in all participants at baseline and 1y follow-up. Multi-MUP analysis and routine EMG will be performed to record and assess MUPs qualitative and semi-quantitatively. Mean duration (simple MUPs), amplitude, and percentage of polyphasic MUPs will be recorded.
Sympathetic skin response in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Sympathetic skin response (SSR) will be conducted to the dominant palm and sole using Sierra Summit EMG system to assess autonomic sympathetic function. The response will be recorded, and the latency determined from the onset of the stimulus artifact to first deflection from baseline. A response will be defined as absent if no reproducible deflection is recorded after consecutive and sporadic stimulations. This test will be performed in post-COVID subjects and age/sex matched controls at baseline and 1y follow-up.
Heart rate variability in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Heart rate variability (HRV) using continuous electrocardiogram (ECG) will be recorded by a two-lead electrocardiograph using the Sierra Summit EMG system. The variation in R-R interval during normal breathing and during deep breathing will be recorded and the variability calculated as maximum heart rate minus minimum heart rate divided by average heart rate, expressed as a percentage. This test will be performed in post-COVID subjects and age/sex matched controls at baseline and 1y follow-up.
Muscle biopsy in the post-COVID subjects and age/sex matched controls | Baseline & 1y follow-up
  Tissue samples of the vastus lateralis muscle will be obtained under local anaesthesia using the percutaneous Bergström technique from the right leg. All muscle samples (~200 mg) will be immediately dissected free of any visible fat, excess blood and connective tissue, and then quickly frozen in liquid nitrogen. Samples were stored at -80°C until the analyses. Muscle biopsies will be collected in post-COVID subjects and age/sex matched controls at baseline and 1y follow-up.
Exercise (in)capacity of post-COVID subjects and age/sex matched controls | Baseline & 48 hours follow-ups of each trial & 1y follow-up
  Cardiopulmonary exercise testing (CPET) will be used to assess exercise capacity as the peak volume of oxygen consumption (VO2 peak) in all participants at several timepoints in this study. First at baseline, then 48h after each exercise trial and finally at the 1y follow-up.
Post-exertional symptoms using the Multifactional Fatigue Inventory (MFI) in post-COVID subjects and age/sex matched controls in response to different exercise trials. | Three exercises trials & 48 hours follow-ups of each trial
  Multifactional Fatigue Inventory (MFI) validated questionnarie will be administrated to assess fatigue exaggeration in response to 3 different exercise trials (high intensity interval training, moderate intensity continuous exercise and strength exercise) between the post-COVID subjects and age/sex matched controls. MFI is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Higher scores reflect higher fatigue levels.
  2 groups x 3 exercise sessions x 3 timepoints per exercise (pre, post and 48h post)
Post-exertional symptoms using the Profile of Mood States (POMS) in post-COVID subjects and age/sex matched controls in response to different exercise trials. | Three exercises trials & 48 hours follow-ups of each trial
  Profile of Mood States (POMS) instrument will be administrated to assess different dimensions of mood states in response to 3 different exercise trials (high intensity interval training, moderate intensity continuous exercise and strength exercise) between the post-COVID subjects and age/sex matched controls. POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment.
  Higher scores reflect increased levels mood states (i.e. higher tension level).
  2 groups x 3 exercise sessions x 3 timepoints per exercise (pre, post and 48h post)
Post-exertional symptoms using the Somatic and Psychological Health REport (SPHERE) instrument in post-COVID subjects and age/sex matched controls in response to different exercise trials. | Three exercises trials & 48 hours follow-ups of each trial
  The Somatic and Psychological HEalth REport (SPHERE) is a 34-item self-report questionnaire that assesses symptoms of mental distress and persistent fatigue. Scores from 12 selected questions will be used to calculate the subscale of SOMA reflect physical fatigue (6 questions) and PHYCH metnal distress (6 questions) respectively. SPHERE instrument will be administrated to assess mental stress and persisent fatigue in response to 3 different exercise trials (high intensity interval training, moderate intensity continuous exercise and strength exercise) between the post-COVID subjects and age/sex matched controls.
  Higher SOMA and PHYCH scores reflect increased levels persistent physical fatigue and mental stress respectively.
  2 groups x 3 exercise sessions x 2 timepoints per exercise (pre and 48h post)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gustafsson, Prof, Study Chair — Karolinska Institutet and Karolinska University Hospital; Helene Rundqvist, PhD, Principal Investigator — Karolinska Institutet; Tommy Lundberg, PhD, Principal Investigator — Karolinska Institutet; Kaveh Pourhamidi, PhD, Study Chair — Karolinska University Hospital; Andrea Tryfonos, PhD, Study Director — Karolinska Institutet
Locations (1):
- Karolinska University Hospital Huddinge, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymised and available in public database and/or as supplementary data in peer reviewed publications following the completion of the study.
Supporting Information: Study Protocol, CSR
Time Frame: Documents will be made available when the summary data are published.

REFERENCES:
- [Derived] Tryfonos A, Jornaker G, Rundqvist H, Pourhamidi K, Melin M, Wallin H, Larsen FJ, Pantelios S, Mutvei AP, Tillander V, Tietge UJF, Diaz SP, Crafoord D, Lovric A, Fernandez-Gonzalo R, Rullman E, Stal P, Gustafsson T, Rundqvist H, Lundberg TR. Muscle Abnormalities in Nonhospitalised Patients With Post-COVID-19 Condition. J Cachexia Sarcopenia Muscle. 2025 Oct;16(5):e70085. doi: 10.1002/jcsm.70085. PMID 41030235
- [Derived] Tryfonos A, Pourhamidi K, Jornaker G, Engvall M, Eriksson L, Elhallos S, Asplund N, Mandic M, Sundblad P, Sepic A, Rullman E, Hyllienmark L, Rundqvist H, Lundberg TR, Gustafsson T. Functional Limitations and Exercise Intolerance in Patients With Post-COVID Condition: A Randomized Crossover Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e244386. doi: 10.1001/jamanetworkopen.2024.4386. PMID 38573638